CLINICAL TRIAL: NCT01524588
Title: C Terminal Peptide Variants of the Fsh Receptor in Women Involved in an Assisted Reproduction Programm : Mechanistic Approach
Brief Title: C Terminal Variants of FSH Receptor
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital, Tours, University Hospital, Tours
Other Study IDs: AOHP07-DR/VARFSHR
Record Dates: First submitted 2011-08-22; First posted 2012-02-02 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Infertility
Keywords: Genotype; Phenotype; Genotypic Variation Between Patients; Genotypic Phenotypic Relationships
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Follicle-stimulating hormone (FSH) is used in medically assisted procreation, to induce an ovarian stimulation in women. However, the FSH dose that has to be injected is quite hard to adjust, because an excess of exogenous hormone could lead to very severe complications for patient. This hormone acts on its cognate receptor, the FSHR, present on the granulosa cells surface, and which regulation involve the intra-cytoplasmic carboxy-terminus domain.

The investigators first aimed to research in the c-terminus part of the receptor the presence of allelic variants that could explain the variations of response to FSH stimulation.

The investigators also would want to complete the data already known on a functionally determinant single nucleotide polymorphism on 680 position in the c-terminus part of the hFSHR.

Then, the investigators would analyze the entire sequence of the hFSHR of patients presenting an unusual phenotype in response to FSH treatment, in order to detect a potential mutation involved in the receptor functionality.

The results of this study could allow us to increase our knowledge on the hFSHR physiology and functionality, in order to adjust treatment to the genetic profile of patients.

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years,
* entering an IVF cycle
* informed consent
* NHS operative

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients involved in an assisted reproduction programm, once engaged in a stimulation protocol
Sampling Method: Non-Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique ROYERE, Principal Investigator — Tours Hospital
Locations (1):
- CHRU de Tours, Tours, France